CLINICAL TRIAL: NCT02727855
Title: Targeted Vaccination of Children in Urban Slums Against Cholera: Evaluation of a Potentially Cost-effective and Impactful Strategy for Deploying Oral Cholera Vaccine in Bangladesh
Brief Title: Cholera Vaccine Investment Strategy in Bangladesh
Acronym: CVIS
Status: Completed | Type: Observational
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Gavi, The Vaccine Alliance (Other); Government of Bangladesh (Other Government)
Responsible Party: Sponsor
Other Study IDs: PR-15091
Record Dates: First submitted 2016-01-16; First posted 2016-04-05 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Cholera
Keywords: Cholera; Vaccine; Strategy
MeSH Terms: conditions — Cholera | interventions — shanchol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Specimens will be preserved for 5 years for future use.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Shanchol — Oral Cholera Vaccine

SUMMARY:
To evaluate the preventive impact, demand, acceptability, uptake, feasibility, and cost-effectiveness of a two-dose regimen of the OCV Shanchol in children living in urban slums in Bangladesh, Investigators will conduct a targeted mass immunization programme, using an innovative approach successfully deployed by the Bangladesh government in its recent countrywide campaign of MR vaccination of 52 million children aged 9 months to 14 years (<15 years). Investigators will undertake a census of a geographic population of approximately 300,000 persons, with GIS locations of each household. This census will be updated every 6 months during the follow-up period to permit tracking of births, deaths, and migrations, including changes in location of each individual's residence. Following the initial census, the OCV will be offered to all non-pregnant individuals aged 1 to 14 years. Operational research and economic studies will evaluate the coverage, feasibility, acceptability, demand, costs and cost-effectiveness of this vaccination programme.

DETAILED DESCRIPTION:
Burden: Cholera remains a major global problem, resulting in more than 100,000 deaths and several million cases annually , mostly children. Vaccination has been reconsidered as a key component of the public health response to cholera. Bangladesh has one of the world's highest burdens of endemic cholera, with an estimated 300,000 cholera cases and over 4,500 deaths annually, and with high caseloads and frequent outbreaks in more than half of the country. The endemicity of cholera in Bangladesh is demonstrated by the predictable yearly occurrence of the disease in the country's high-risk districts and the repetitive seasonal pattern of cholera outbreaks, either in spring or autumn, or both .

Knowledge gap: More evidence is needed to address uncertainties around the cholera disease burden, as well as the impact, feasibility, and cost-effectiveness of various vaccination strategies against cholera, to add to the existing knowledge base. A special need for acquiring field evidence of these vaccine attributes in settings with endemic cholera, which account for a very large fraction of the global cholera disease burden, is also recognized .

Relevance: Nonetheless, the assertion that selective vaccination of children with OCV is an impactful approach to controlling cholera at the population level rests on unproven assumptions, since there are no studies that directly address this vaccination strategy. Therefore, further study on whether targeted mass immunization can create efficiencies that general mass immunization would not, is warranted. The Investigators therefore believe that the most compelling question for the control of endemic cholera in Bangladesh is how targeting 1-14 year olds in urban slums, using the established platform of targeted mass childhood immunization recently deployed by the GOB for measles-rubella (MR) vaccine, impacts on the overall burden of cholera in the population and how feasible and cost-effective this strategy is. Addressing these questions will add to the evidence base on the most cost efficient and effective settings and strategies for use of OCV to control endemic disease and optimize health impact.

Hypothesis : Vaccination of children under 15 years of age in urban slums of Dhaka will confer at least 50% overall protection to the entire population through combined direct and indirect protective effects and it will be cost effective.

Objectives:To evaluate the feasibility, efficiency, and impact of a two-dose regimen of the oral cholera vaccine (OCV) Shanchol delivered to children aged 1-14 years residing in urban slums, leveraging a targeted mass immunization delivery platform used for other vaccines in Bangladesh.

Methods: Observational design based on the contrast of persons who do and do not get vaccinated according to public health practice(Age-targeted mass immunization program).

ELIGIBILITY:
Inclusion Criteria:

* All healthy, consenting, non-pregnant (as ascertained by history) residents of a high risk group, 1 to 14 years of age, of the study area will be included in the study.

Exclusion Criteria:

* Aged less than 1 year and more than 14 years
* History of intake of any cholera vaccine
* Pregnant women (identified through verbal screening)

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will be recruited from different wards of Dhaka city corporation (wards 42, 43, 45, 46, 47, 48, 58, 91 and 92 which are now numbered as 29,30,32,33,34 of Dhaka North City Corporation and 14,22,55,56,57 of Dhaka South City Corporation respectively).
Sampling Method: Probability Sample
Enrollment: 75170 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with two doses of oral cholera vaccine (Shanchol) will get protection | 2 years from dosing
  Shanchol vaccine will be given to healthy , non pregnant residents aged 1-14 years in Dhaka, Bangladesh against culture proven vibrio cholerae O1 diarrhoea which has been detected in all treatment settings serving the catchment population.

SECONDARY OUTCOMES:
Cholera vaccine coverage | 10 months
  Vaccination status of children by age, sex, socioeconomic characteristics of the household evaluation
Vaccine acceptability | 17 months
  Exit interviews with caregivers, direct observation of vaccination sessions, in-depth interviews and focus groups with guardians of vaccine recipients and of children not receiving vaccine will be conducted using qualitative guidelines to evaluate the taste of the vaccine, the convenience of the vaccine delivery program, willingness to participate in similar future vaccination programmes,general concerns about the vaccine and the vaccine program
Vaccine feasibility | 17 months
  Quantitative survey with a structured questionnaire administered to vaccination team members, and in depth interviews of purposefully selected vaccine supervisors and programme managers and focus group discussions with vaccination teams to evaluate the barriers faced in implementing the programme, availability of infrastructural supports, logistics and human resources, the adequacy of the vaccine transportation system, adequacy of cold chain and vaccine storage management, suitability of vaccination session management
Incidence of cholera among vaccinated individuals in vaccination area | Two years after completion of vaccination
  Vaccine induced protective immunity and the indirect protection ( Herd immunity) will be estimated from comparing the incidence of cholera among vaccine recipients in the vaccination area and the incidence of cholera among vaccine non recipients in the same area.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Firdausi Qadri, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to anybody.

REFERENCES:
- [Result] Ali M, Lopez AL, You YA, Kim YE, Sah B, Maskery B, Clemens J. The global burden of cholera. Bull World Health Organ. 2012 Mar 1;90(3):209-218A. doi: 10.2471/BLT.11.093427. Epub 2012 Jan 24. PMID 22461716
- [Result] Sur D, Lopez AL, Kanungo S, Paisley A, Manna B, Ali M, Niyogi SK, Park JK, Sarkar B, Puri MK, Kim DR, Deen JL, Holmgren J, Carbis R, Rao R, Nguyen TV, Donner A, Ganguly NK, Nair GB, Bhattacharya SK, Clemens JD. Efficacy and safety of a modified killed-whole-cell oral cholera vaccine in India: an interim analysis of a cluster-randomised, double-blind, placebo-controlled trial. Lancet. 2009 Nov 14;374(9702):1694-702. doi: 10.1016/S0140-6736(09)61297-6. Epub 2009 Oct 8. PMID 19819004
- [Result] Glass RI, Becker S, Huq MI, Stoll BJ, Khan MU, Merson MH, Lee JV, Black RE. Endemic cholera in rural Bangladesh, 1966-1980. Am J Epidemiol. 1982 Dec;116(6):959-70. doi: 10.1093/oxfordjournals.aje.a113498. PMID 7148820